CLINICAL TRIAL: NCT01005602
Title: Use of a Simplified Nomogram and Pharmacogenetics to Individualize Digoxin Dosing in Heart Failure Patients vs. Standard Care
Brief Title: Digoxin Dosing in Heart Failure: A Simplified Nomogram Versus Standard Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Principal Investigator, Robert J. DiDomenico, Clinical Associate Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCP 2006-07; 2008-05762
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: Digoxin; Pharmacokinetics; Dosing; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digoxin Dosing per Nomogram (Experimental): Subjects will have their digoxin maintenance dose determined according to the nomogram we have developed.
  Interventions: Other: Digoxin Dosing per Nomogram; Drug: Digoxin
- Standard Digoxin Dosing (Other): This arm represents historical control subjects in whom the dose of digoxin was determined at the physician's discretion using traditional dosing methods.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Other: Digoxin Dosing per Nomogram — Simplified dosing nomogram for digoxin. The dose is determined by plotting a subject's creatinine clearance (x-axis) and ideal body weight (y-axis) on the nomogram. Alternatively, the dose may be determined by plotting creatinine clearance (x-axis) and gender/height (z-axis).
  Arms: Digoxin Dosing per Nomogram
Drug: Digoxin — All patients included in the trial were treated with digoxin as clinically indicated. The intervention for this study required determining the digoxin dose via a proposed nomogram.
  Other Names: Lanoxin

SUMMARY:
Dosing methods for digoxin, a drug used to treat heart failure, have not been updated in decades despite evidence in recent years suggesting that blood levels of digoxin achieved with traditional dosing practices may increase the risk of adverse events. We developed a simple dosing tool that targets lower blood levels of digoxin that have been associated with improved outcomes compared to higher blood levels. The aim of this study is to determine if this simplified dosing tool is more effective than standard digoxin dosing practices at achieving lower blood levels and also to determine if digoxin dosing may be further optimized by incorporating patients' genetic information believed to influence the drug's properties.

DETAILED DESCRIPTION:
Digoxin is recommended as adjunctive therapy in patients with left ventricular dysfunction and symptoms of heart failure despite treatment with standard therapy. Recently, the therapeutic range for digoxin in patients with heart failure has been redefined to a narrower therapeutic window (0.5 - 0.9 ng/ml) because lower serum levels in this range have been associated with improved survival whereas higher serum levels have been associated with increased mortality. However, dosing methods have not been updated to reflect the newly defined therapeutic range for digoxin. We developed a simplified dosing nomogram for digoxin in patients with heart failure designed to achieve serum digoxin concentrations (SDC) within the new therapeutic range using retrospective data. The long-term goal of this study is to prospectively validate the ability of our digoxin dosing nomogram to achieve desired SDC and provide clinicians a simplified tool to optimize digoxin dosing in patients with heart failure. Because digoxin is a substrate of the efflux pump p-glycoprotein (pGP) and genetic polymorphisms of the MDR1 gene (known to regulate pGP expression) have demonstrated conflicting results on the pharmacokinetic profile of digoxin, we will also characterize the influence MDR1 functional gene variants may have on digoxin dosing. This study will include a total of 170 subjects with symptomatic heart failure treated with digoxin, comparing steady-state SDC in a prospective group of patients dosed according to our nomogram to a historical control group in whom the dose of digoxin was derived from standard dosing practices. We will also conduct an analysis of genetic polymorphisms of the MDR1 gene known to affect digoxin pharmacokinetics. The primary objectives of the study are to compare the percentage of patients in each group achieving steady-state SDC within the desired range of 0.5 - 0.9 ng/ml, characterize the relationship between genetic variability in the MDR1 gene and digoxin dosing, and to update our digoxin dosing nomogram to account for the clinical and genetic variability shown to have the greatest influence on digoxin dosing. The rationale for this study is that lower doses of digoxin are recommended because lower SDC are associated with improved survival. Therefore, digoxin dosing methods must be updated to reflect these recommendations and account for genetic variability of the MDR1 gene in an effort to improve clinical outcomes and minimize the potential for adverse events. To address these issues, the specific aims of this research are:

Aim 1: Compare steady-state SDC observed using our dosing nomogram to those obtained using standard dosing practices.

Aim 2: Characterize the relationship of the genetic variability of the MDR1 gene and SDC observed using our digoxin dosing nomogram.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Diagnosis of heart failure secondary to left ventricular dysfunction
* Receiving chronic digoxin therapy or digoxin therapy is being initiated

Exclusion Criteria:

* Pregnant
* Unstable renal function, defined as either a rise in serum creatinine by > 0.5mg/dl from baseline or a decrease in creatinine clearance by 25% or more within two to four weeks of study entry.
* End-stage renal disease requiring hemodialysis
* Concomitant therapy with drugs known to interact with digoxin (e.g., amiodarone, quinidine, verapamil, macrolide antibiotics)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J DiDomenico, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Bauman JL, DiDomenico RJ, Viana M, Fitch M. A method of determining the dose of digoxin for heart failure in the modern era. Arch Intern Med. 2006 Dec 11-25;166(22):2539-45. doi: 10.1001/archinte.166.22.2539. PMID 17159022
- [Derived] DiDomenico RJ, Bress AP, Na-Thalang K, Tsao YY, Groo VL, Deyo KL, Patel SR, Bishop JR, Bauman JL. Use of a simplified nomogram to individualize digoxin dosing versus standard dosing practices in patients with heart failure. Pharmacotherapy. 2014 Nov;34(11):1121-31. doi: 10.1002/phar.1480. Epub 2014 Aug 28. PMID 25164709

RESULTS

PARTICIPANT FLOW:
Groups:
- Digoxin Dosing Per Nomogram: Subjects will have their digoxin maintenance dose determined according to the nomogram we have developed.
  Dosing nomogram for digoxin: Simplified dosing nomogram for digoxin. The dose is determined by plotting a subject's creatinine clearance (x-axis) and ideal body weight (y-axis) on the nomogram. Alternatively, the dose may be determined by plotting creatinine clearance (x-axis) and gender/height (z-axis).
Period: Overall Study
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing
Started | 66 | 66
Completed | 65 (One patient completed the trial but was excluded from data analyses due to unreliable clinical data.) | 66
Not Completed | 1 | 0
Not completed — Excluded due to unreliable clinical data | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15) | 63 (15) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 63
  Male | 38 | 30 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 40 | 86
  White | 7 | 15 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 11 | 23
Ideal body weight [Mean (Standard Deviation); unit: kg] — Ideal body weight (IBW) as determined by the method of Devine. (Devine BJ. Drug Intell Clin Pharm 1974;8:650-5.)
  kg | 67 (10) | 62 (11) | 65 (11)
Total body weight [Mean (Standard Deviation); unit: kg] | 100 (34) | 85 (27) | 92 (32)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (10.4) | 29.9 (8.9) | 31.6 (9.8)
Creatinine clearance [Mean (Standard Deviation); unit: ml/min] | 66 (10) | 51 (22) | 58 (25)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 71 (22) | 59 (23) | 65 (23)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving a Desired Steady-state Serum Digoxin Concentration Between 0.5 - 0.9ng/ml
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Number; unit: percentage of participants
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing
Number analyzed (Participants) | 65 | 66
percentage of participants | 38.5 | 34.8

2. Secondary Outcome: Mean Serum Digoxin Concentration
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing
Number analyzed (Participants) | 65 | 66
ng/ml | 0.52 (0.30) | 1.12 (0.58)

3. Secondary Outcome: Serum Digoxin Concentration < 1.0 ng/ml
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Number; unit: percentage of participants
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing
Number analyzed (Participants) | 65 | 66
percentage of participants | 86.2 | 42.4

4. Secondary Outcome: Serum Digoxin Concentration by ABCB1 Single Nucleotide Polymorphism (SNP) C1236T
Description: 55 patients in the Digoxin Dosing per Nomogram group consented to the Pharmacogenetic substudy and provided blood samples to perform pharmacogenetic analyses. We compared serum digoxin concentrations by ABCB1 genotype.
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Wild Type: Genotypes for the ABCB1 single nucleotide polymorphism C1236T
Arm/Group | Wild Type | CT Genotype | TT Genotype
Number analyzed (Participants) | 31 | 20 | 4
ng/ml | 0.52 (0.27) | 0.56 (0.37) | 0.58 (0.29)

5. Secondary Outcome: Serum Digoxin Concentration by ABCB1 SNP C3435T
Description: Serum digoxin concentration by genotypes for the ABCB1 SNP C3435T
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Wild Type (CC) | CT Genotype | TT Genotype
Number analyzed (Participants) | 27 | 25 | 3
ng/ml | 0.54 (0.28) | 0.54 (0.35) | 0.46 (0.07)

6. Secondary Outcome: Serum Digoxin Concentration by ABCB1 SNP G2677T/A
Description: Serum digoxin concentration by ABCB1 SNP genotypes
Time Frame: Steady-state (2 - 4 weeks after initiation)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Wild Type (GG) | GT Genotype | TT Genotype | GA Genotype
Number analyzed (Participants) | 38 | 12 | 3 | 2
ng/ml | 0.54 (0.27) | 0.50 (0.42) | 0.66 (0.30) | 0.40 (0.13)

ADVERSE EVENTS:
Arm/Group | Digoxin Dosing Per Nomogram | Standard Digoxin Dosing
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 0/65 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No